CLINICAL TRIAL: NCT00150488
Title: URACYST® For the Treatment of GAG Deficient Interstitial Cystitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. J. Curtis Nickel (Other)
Collaborators: Stellar Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Dr. J. Curtis Nickel, Principal Investigator, Queen's University
Organization: Queen's University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uracyst-Stellar
Record Dates: First submitted 2005-09-06; First posted 2005-09-08 (Estimated); Results first posted 2023-07-27 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2022-09

CONDITIONS: Painful Bladder Syndrome; Interstitial Cystitis
Keywords: PBS; Painful Bladder Syndrome; Interstitial Cystitis; chrondroitin sulfate
MeSH Terms: conditions — Cystitis, Interstitial

STUDY DESIGN:
Intervention Model Description: Uracyst
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Uracyst® single arm open label Treatment Group
  Interventions: Device: Uracyst

INTERVENTIONS:
Device: Uracyst — 2% weekly for 6 weeks, monthly for 4 months
  Other Names: chondroitin sulphate

SUMMARY:
This protocol describes a multi-centre, community based open label study designed to assess the efficacy and safety of intravesical sodium chrondroitin sulfate (Uracyst®) in the treatment of patients with a clinical diagnosis of interstitial cystitis (IC).

The safety of the study product will be evaluated through the incidence of adverse events and from results of physical examinations and laboratory tests.

DETAILED DESCRIPTION:
The primary efficacy endpoint will be the percent responders to treatment as indicated by improvement on a seven-point Patient Global Assessment scale at week 10 (after 6 treatments) compared to baseline. The patient evaluates the overall change in their condition as markedly improved, moderately improved, slightly improved, no change, slightly worse, moderately worse or markedly worse.

Secondary efficacy objectives will be as follows:

1. Improvement in individual IC symptoms during the treatment period and at week 10 (after 6 treatments) compared to baseline.

   Pain and urgency scores (0-10 cm VAS) will be obtained using patient on-site questionnaires prior to first treatment (baseline), and again for weeks 4, 6, 10, 14, 18, 22 and 24.
2. Change in Patient Symptom/Problem Index scores over the course of the treatment until the end of study (week 24) compared to baseline.

   The validated O'Leary Symptom Problem/Index will be completed prior to first treatment (baseline) and again for weeks 4, 6, 10, 14, 18, 22 and 24.

   The validated PUF questionnaire will be completed prior to first treatment (baseline) and again for weeks 4, 6, 10, 14, 18, 22 and 24.
3. Change in patient condition every month throughout the therapy and treatment follow-up.

In addition to measuring the change in patient condition at week 14, the Patient Global Assessment will be completed at weeks 4, 6, 10, 14, 18, 22 and 24.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following eligibility criteria in order to be enrolled in this study.

1. Clinical diagnosis of interstitial cystitis
2. Legally majority female capable and willing to provide informed consent
3. Negative blood test for pregnancy at baseline or assurance of previous surgery, condition or state rendering conception impossible
4. A sterile bacterial urine culture no more than thirty (30) days prior to first treatment
5. An average urinary frequency of at least 11 times per 24-hour day
6. An average pain/discomfort score of 4 or greater on a 0-10cm VAS scale
7. Available for the duration of the study including treatment and follow-up (4 months)

Exclusion Criteria:

1. Pregnant or lactating
2. Currently receiving or having received investigational drugs thirty (30) days or less prior to screening
3. Currently receiving or having had prior therapy with intravesical treatment (eg. Uracyst, Cystistat®, heparin or BCG)
4. Receiving therapy for less than three months with antidepressants, antihistaminics, hormonal agonists or antagonists; hence patient not stabilized on therapy. (Stable therapy defined as continuous treatment for at least three months.)
5. Currently receiving or having received prior therapy with oral pentosanpolysulfate (Elmiron) 3 months or less prior to screening
6. IC symptoms relieved by antimicrobials, anticholinergics or antispasmodics
7. Bladder capacity of greater than 500 ml on awake cystometry using liquid filling medium
8. Neurologic disease affecting bladder function; any previous surgery or procedure having affected bladder function
9. Current urinary tract infection (must be treated and have a negative culture before study entry)
10. Current diagnosis of chemical, tuberculous or radiation cystitis
11. History of bladder or lower ureteral calculi
12. History of cancer within the last five years other than adequately treated non-melanoma skin cancers
13. Active sexual transmitted disease
14. Current vaginitis
15. Endometriosis
16. Any condition/disease which in the opinion of the investigator could interfere with patient compliance and/ or interfere with the interpretation of the treatment results

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-09; Primary Completion 2008-01 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Curtis Nickel, MD FRCSC, Principal Investigator — Queen's University
Locations (1):
- Centre for Advanced Urological Research, Kingston General Hospital, Kingston, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Uracyst Treatment Group: Moderately/severely symptomatic Interstitial cystitis patients
Period: Overall Study
Arm/Group | Uracyst Treatment Group
Started | 53
Completed | 53
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Uracyst Treatment Group: Subjects with diagnosis of Interstitial Cystitis with positive potassium sensitivity test
Arm/Group | Uracyst Treatment Group
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 52
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 53
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Canada | 53

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Responders to Treatment
Description: indicated by a marked or moderate improvement on a seven-point patient Global Response Assessment (GRA) scale compared with baseline
Time Frame: Week 10 (4 weeks after the initial six treatments
Measure: Count of Participants; unit: Participants
Arm/Group | Uracyst Treatment Group
Number analyzed (Participants) | 53
Participants | 25

2. Secondary Outcome: Change in Likert Pain Score From Baseline at 10 Weeks
Description: Scale of 0-10; subjects report 0=no pain and 10 pain as bad as you can imagine.
Time Frame: Baseline and 10 Weeks
Measure: Mean (Standard Deviation); unit: units on a scale 0-10
Groups:
- Uracyst Treatment Group: The cohort of interstitial cystitis patients in this trial was chronic, moderately to severely symptomatic and comparable with those enrolled in recent intravesical therapy treatment trials.
Arm/Group | Uracyst Treatment Group
Number analyzed (Participants) | 53
units on a scale 0-10 | -2.6 (1.5)
Statistical Analysis 1: Comparison: Uracyst Treatment Group; Test type: Other — Compared to baseline; p < 0.001, Chi-squared

ADVERSE EVENTS:
Time Frame: 4 months
Groups:
- Uracyst Treatment Goup: Uracyst®
  Uracyst: 2% weekly for 6 weeks, monthly for 4 months
Arm/Group | Uracyst Treatment Goup
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 28/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Uracyst Treatment Goup (N=53)
Upper respiratory (Respiratory, thoracic and mediastinal disorders) | 19 (19)
unrelated pain (Nervous system disorders) | 17 (17) — pain unrelated to bladder
Genital burning/discomfort (Skin and subcutaneous tissue disorders) | 10 (10)
Urinary Tract Infection (Infections and infestations) | 6 (6)
Gastro intestinal (Gastrointestinal disorders) | 6 (6)
Increased bladder symptoms (urgency, frequency, incontinence (Renal and urinary disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No